CLINICAL TRIAL: NCT01831713
Title: Evaluation of Pulmonary Blood Flow Patterns Using Transthoracic Doppler in Patients With Congestive Heart Failure
Brief Title: Pulmonary Blood Flow Measurements in CHF Patients
Status: Terminated | Type: Observational
Why Stopped: Changing staff
Sponsor: Echosense Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIH DOP08
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2012-08

CONDITIONS: Congestive Heart Failure (CHF)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CHF patients and Controls: CHF patients refer to Decompensated patients and Compensated patients

SUMMARY:
Historically, transthoracic Doppler echocardiography has been unable to provide interpretable data of blood flow within the lung parenchyma because of air attenuation of Doppler signals. Recently, a transthoracic Doppler system known as the Sonara/tek Transcranial Doppler (TCD) System has been developed that can identify parenchymal pulmonary blood flow (PPBF) signals. The ability to non-invasively collect information regarding the pulmonary aspect of the cardio-pulmonary system may provide valuable information and new insights into the structural and functional characteristics of the lung parenchyma and vasculature in health and disease states.

DETAILED DESCRIPTION:
This new system was previously studied among 31 healthy volunteers and one subject with atrial fibrillation.1 Pulsed spectral Doppler signals were obtained over the chest wall using a signal processing and algorithm package in conjunction with a non-imaging Doppler device coupled with an electrocardiogram. Clear reproducible lung Doppler signals (LDS) originating from different elements and phases of cardiac activity that generate mechanical waves which propagate throughout the lung were expressed in pulsatile changes in ultrasound reflections.

After the completion of the first 25 patients in our pilot study, we have received some valuable information. After assessing patients with CHF and pulmonary hypertension, we identified signals particular to the CHF group. There were unique features that were never observed in the normal patients. On top of the regular Lung Doppler signals seen in normal patients, high velocity "disorganized" variable signals that were not synchronous with the heart beat, but rather sometimes with respiration were observed. We believe that the signals may represent popping open of small bronchi surrounded by "water filled" parenchyma. These events that generate very strong reflector like signals may represent the movement of fluid at the blood vessel-alveolar air junction.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  1. Age over 50 years
  2. Belongs to one of the following categories:

     A. Decompensated CHF: patients with overt pulmonary congestion or pulmonary edema on admission, evident both clinically and by chest x-ray. Patients may be with or without a Swan-Ganz catheter.

     B. Compensated CHF: patients with significant CHF (NYHA II-IV) who are well controlled and without evidence of pulmonary congestion or pulmonary edema on admission.

     C. Non-CHF controls: patients without CHF and without any of the following: pulmonary hypertension, any known pulmonary disease, uncontrolled hypertension.
  3. Signed Informed Consent

Exclusion Criteria:

* Chronic obstructive pulmonary disease (COPD) Asthma Interstitial lung disease Any other obstructive or restrictive lung diseases Pneumonia- currently or in the past 3 months prior to inclusion Current or past pulmonary embolism Non-cardiogenic pulmonary edema or lung injury (e.g. ARDS) Right sided pleural effusion that is not mild Severe kyphosis, scoliosis or chest wall deformity

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CHF patients admitted to the cardiology telemetry unit and to the CCU
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Diagnose specific patterns of doppler signals in CHF patients | December 2013

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Chen, MD, Study Director — Lenox Hill Hospital, 100East 77 Street New York, NY 10075
Locations (1):
- NSLIJ Lenox Hill hospital, 100East 77 Street, New York, New York, United States